CLINICAL TRIAL: NCT00898612
Title: Using the Transcriptome for Early Detection of Graft Versus Host Disease in Allogeneic Bone Marrow Transplantation
Brief Title: Early Detection of Graft-Versus-Host Disease in Patients Undergoing a Donor Bone Marrow Transplant
Status: Withdrawn | Type: Observational
Why Stopped: No Patients enrolled
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Roberta H. Adams, M.D., Mayo Clinic Cancer Center
Other Study IDs: CDR0000588925; P30CA015083 (NIH); 878-05 (Other: Mayo Clinic Cancer Center); 878-05 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Lymphoma
Keywords: stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; juvenile myelomonocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; childhood myelodysplastic syndromes; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; myelodysplastic/myeloproliferative neoplasm, unclassifiable; poor prognosis metastatic gestational trophoblastic tumor; previously treated childhood rhabdomyosarcoma; previously treated myelodysplastic syndromes; recurrent Wilms tumor and other childhood kidney tumors; recurrent childhood rhabdomyosarcoma; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent malignant testicular germ cell tumor; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; refractory multiple myeloma
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Recurrence; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myeloid, Acute; Leukemia, Hairy Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Myeloproliferative Disorders; Wilms Tumor; Neuroblastoma; Carcinoma, Ovarian Epithelial; Testicular Neoplasms; Multiple Myeloma; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients who have undergone a donor bone marrow transplant may help doctors learn more about changes that occur in DNA and identify biomarkers related to graft-versus-host disease. It may also help doctors predict how patients will respond to a donor bone marrow transplant.

PURPOSE: This laboratory study is looking at early detection of graft-versus-host disease in patients undergoing a donor bone marrow transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify detectable changes in the transcriptomic or proteomic expression prior to clinical manifestations of graft-versus-host disease (GVHD) in blood samples from at-risk patients who have undergone allogeneic bone marrow transplantation.

Secondary

* Characterize changes in the transcriptome or proteome expression pattern which are predictive of clinically significant GVHD in these patients.
* Develop reliable tests which enable early intervention for these patients.

OUTLINE: Blood samples are collected prior to and just after typical onset of clinical graft-vs-host disease (GVHD) on days 1, 7-10, 20-23, 30-33, and 60 after allogeneic bone marrow transplantation. RNA is quantified and assessed by microarray analysis to identify changes to transcriptome or proteome expression and markers predictive of the onset of clinical GVHD. Samples are also stored for future analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Any patient undergoing an allogeneic bone marrow transplantation at one of the participating Mayo Clinic sites

PATIENT CHARACTERISTICS:

* Body weight ≥ 15 kg
* Not pregnant
* Not a prisoner

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing allogeneic bone marrow transplantation at participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Identification of changes in the transcriptome or proteome expression prior to clinical manifestations of graft-versus-host disease (GVHD) in patient blood samples | Patients beyond period of risk for developing acute GVHD
  Once a minimum of 20 patients have been enrolled and clinically are beyond their period of risk of developing acute GVHD, samples from at least 5 patients who have developed acute GVHD are compared to samples from at least 5 patients who have had no detectable clinical GVHD. If no differences are detected, additional patients/samples will be enrolled/analyzed.

SECONDARY OUTCOMES:
Characterization of changes in the expression patterns which are predictive of clinically significant GVHD | Patient beyond period of risk for developing acute GVHD
Development of reliable tests to predict GVHD in time for early intervention | Patient beyond period of risk for developing acute GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Adams, MD, Principal Investigator — Mayo Clinic Hospital
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States